CLINICAL TRIAL: NCT00051233
Title: Schizophrenia Patient and Family Continuity of Care
Brief Title: Treatment of Schizophrenia Through Internet-Based Psychoeducation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH063484 (NIH); R01MH063484 (NIH); DSIR SE-DR
Record Dates: First submitted 2003-01-07; First posted 2003-01-08 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

INTERVENTIONS:
Procedure: World Wide Web-Based Psychoeducation

SUMMARY:
The purpose of this study is to assess the effectiveness of a Web-based psychoeducational program in helping people with schizophrenia and their families manage the disease.

DETAILED DESCRIPTION:
This study will provide a comprehensive psychoeducational program which includes education, social support, information, coping strategies, and guidance from mental health, social services, and medical professionals. This study will work to reduce relapse, facilitate patient rehabilitation, decrease family distress, and improve family well being.

Patients and their families participate in an in-person Psychoeducational Survival Skills Workshop that is designed to provide patients and their families with basic information about schizophrenia and its treatment. After the workshop, participants are provided with 6 Web-based modules that are designed to increase mental health and schizophrenia knowledge. Patient relapse, family distress, family knowledge of schizophrenia, and data on user's acceptance and utilization are measured to determine the intervention's effectiveness.

ELIGIBILITY:
Inclusion Criteria

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder
* At least 4 hours/week in-person contact with a family member
* Primary caregiver with a telephone
* Patient and primary caregiver speak and read English

Exclusion Criteria:

* Enrolled in another clinical trial
* Evidence of organic brain syndrome
* Current alcohol or substance abuse that could explain the presenting index psychotic episode
* DSM-IV diagnosis of psychoactive substance dependency

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2003-01; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Overall Officials: Armando J Rotondi, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States